CLINICAL TRIAL: NCT00169221
Title: CARISSA Trial - Multicenter Randomized Phase II Trial Comparing Post-operative Radiotherapy and Cisplatin Alone or in Combination With the EGFR Inhibitor ZD 1839 (Iressa) in Upper Aerodigestive Tract Carcinomas
Brief Title: Post-operative Radiotherapy With Cisplatin Alone or in Combination With Iressa in Upper Aerodigestive Tract Carcinomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Toxicity in an independent study IMEX. The trial was subsequently terminated (54 pts instead of 140) despite safety analyses showing no excess of toxicity
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2004-02
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-11-15 (Estimated); Status verified 2011-11

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Gefitinib; Chemoradiotherapy; Cisplatin

ARMS (2):
- postop chemoradio with cisplatin (Active Comparator): postoperative chemoradiotherapy with cisplatin
  Interventions: Radiation: chemoradiotherapy with cisplatin
- postop chemoradio (cisplatin)+gefitinib (Experimental): postoperative chemoradiotherapy with cisplatin + gefitinib
  Interventions: Drug: Iressa (Gefitinib)

INTERVENTIONS:
Drug: Iressa (Gefitinib) — postoperative chemoradiotherapy with cisplatin + gefitinib
  Arms: postop chemoradio (cisplatin)+gefitinib
Radiation: chemoradiotherapy with cisplatin — postoperative chemoradiotherapy with cisplatin
  Arms: postop chemoradio with cisplatin

SUMMARY:
This trial will be an open multicentric randomized phase II study comparing post-operative radiotherapy + cisplatin associated or not with Iressa in upper aerodigestive tract carcinomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients with upper aerodigestive tract carcinomas (all sites included) having surgical resection and eligible for post-operative radiation + cisplatin.
* Patient having a tumoral biopsy (0.5 - 1 cm3) stored in liquid nitrogen at time of surgical resection (patients with small tumors located in larynx for instance will not be included)
* Patients receiving post-operative radiation (>=60 Gy on tumor bed and/or cervical area), associated with cisplatin, 6 weeks after surgery at the latest.

Exclusion Criteria:

* previous history of cancer (except skin basal cell carcinoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2005-09; Primary Completion 2009-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Rene-Jean Bensadoun, MD, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, France

REFERENCES:
- [Derived] Thariat J, Bensadoun RJ, Etienne-Grimaldi MC, Grall D, Penault-Llorca F, Dassonville O, Bertucci F, Cayre A, De Raucourt D, Geoffrois L, Finetti P, Giraud P, Racadot S, Moriniere S, Sudaka A, Van Obberghen-Schilling E, Milano G. Contrasted outcomes to gefitinib on tumoral IGF1R expression in head and neck cancer patients receiving postoperative chemoradiation (GORTEC trial 2004-02). Clin Cancer Res. 2012 Sep 15;18(18):5123-33. doi: 10.1158/1078-0432.CCR-12-1518. Epub 2012 Aug 1. PMID 22855581